CLINICAL TRIAL: NCT04067622
Title: Novel Arm Restraint For Critically Ill Patients To Reduce Immobility, Sedation, Agitation and Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Johns Hopkins University (Other); University of California, San Diego (Other); Healthy Design, LLC (Unknown)
Responsible Party: Principal Investigator, Renee Stapleton, Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS-18-0353
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Acute Respiratory Failure; Encephalopathy; ARDS; Sepsis; Critical Illness
MeSH Terms: conditions — Brain Diseases; Sepsis; Critical Illness

STUDY DESIGN:
Intervention Model Description: Within-patient, randomized crossover design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exersides restraints first (Other): Patients in this arm will wear the novel Exersides restraint during hours 1-4 on Day 1, then switched to soft wrist restrains during hours 5-8. On Day 2, patients in this arm will will wear soft wrist restraints during hours 1-4, and Exersides during hours 5-8. They will then wear Exersides during study days 3-6.
  Interventions: Device: Exersides
- Traditional restraints first (Other): Patients in this arm will wear soft wrist restraints during hours 1-4 on Day 1; they will then be switched to the novel Exersides restraint during hours 5-8. On Day 2, patients in this arm will will wear Exersides during hours 1-4, and soft wrist restraints during hours 5-8. They will then wear soft wrist restraints during study days 3-6.
  Interventions: Device: Exersides

INTERVENTIONS:
Device: Exersides — A novel arm restraint which permits arm mobility but prohibits hands from reaching oral/nasal endotracheal and feeding tubes or intravenous lines.

SUMMARY:
This study evaluates a novel arm restraint compared with traditional soft wrist restraints in older critically ill patients. The primary outcome is upper extremity mobility measured by actigraphy, and secondary outcomes include sedation, agitation, satisfaction, and acceptability.

DETAILED DESCRIPTION:
The goal of this Fast-Track STTR project is to optimize and test a novel arm restraint in older critically ill patients that increases mobility; reduces agitation, use of sedative medications, and delirium; and exhibits high satisfaction and acceptability among hospital staff, family members, and patients. Older critically ill patients are often immobilized with wrist restraints to prevent self-removal of tubes and lines and are sedated to reduce agitation caused by their restraints and endotracheal (breathing) tube. This sedation and immobility lead to complications, including delirium and muscle weakness, that are independently associated with long term cognitive impairment, reduced physical functioning, and mortality. Specifically, the incidence and duration of delirium in the ICU are strongly and independently associated with long-term cognitive impairment that is similar to Alzheimer's Disease and Related Dementias.

Healthy Design is developing the novel ExersidesTM restraint that allows arm mobility but prohibits hands from reaching oral/nasal endotracheal and feeding tubes or intravenous lines. Because it permits mobility, ExersidesTM may reduce agitation and the need for sedatives. In preliminary pilot testing, ExersidesTM has demonstrated very encouraging results. The objectives of this STTR Fast-Track project are to optimize ExersidesTM and evaluate it in a randomized controlled trial (RCT) in older critically ill patients at high risk for delirium and associated long-term cognitive impairment. The multidisciplinary investigator team has expertise in critical care, extensive experience in conducting ICU RCTs, and a history of successful collaboration.

Phase I of the STTR, during which the novel restraint device was modified based on feedback from healthy volunteers and a single-center prospective pilot study was performed in 8 older patients with acute respiratory failure, has already been completed. The Phase I pilot study has demonstrated that 1) the revised ExersidesTM prototype is safe and 2) the RCT proposed in Phase II is feasible.

Therefore, Phase II of the STTR will now occur. In Phase II, a multi-site within-patient crossover RCT in older critically ill patients requiring restraint will be conducted to test the following outcomes in ExersidesTM versus traditional wrist restraint: 1) Mobility assessed by actigraphy (primary outcome); 2) Agitation, delirium, and medication use (secondary outcomes); and 3) Satisfaction with and acceptability/perceptions of the device (secondary outcomes). Successful completion of this project will result in an ExersidesTM restraint that is ready for final optimization in preparation for commercialization, and is suitable for larger clinical studies to demonstrate effectiveness reducing long-term cognitive impairment in older ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Requiring ICU care
* Requiring wrist or mitt restraints and has active physician order
* Expected ICU stay ≥2 days after enrollment
* Responsive to verbal stimulus

Exclusion Criteria:

* Bilateral upper extremity impairments (e.g. arm injuries) or problems (e.g. severe skin breakdown) that prevent use of novel restraint device. Normal use of one arm (e.g. unilateral upper extremity amputation) is acceptable.
* Very limited mobility of bilateral upper extremities prior to admission (e.g. bilateral frozen shoulders). Normal use of one arm is acceptable.
* Pre-existing severe neuromuscular condition inhibiting or axacerbating upper extremity movement (e.g. Guillain-Barre, severe tremor, myoclonus)
* Neuromuscular blocker infusion (eligible once infusion discontinued if other inclusion criteria met)
* Pre-existing severe cognitive impairment or language barrier prohibiting outcome assessment
* Expected death or withdrawal of life-sustaining treatments within 6 days from enrollment
* Incarcerated
* Pregnant
* Attending physician declines patient enrollment
* LAR unavailable to consent (and patient is unable to consent)
* Patient or LAR decline consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Mobility assessed by actigraphy | Up to 6 days
  Upper extremity mobility will be evaluated by actigraphy. The Philips Respironics Spectrum Plus® actigraph is a commercially-available actigraphy device weighing 16 grams. It contains a battery-powered activity monitor and uses a highly sensitive accelerometer to monitor the occurrence and degree of motion. Only patients who wear both the novel restraint and traditional soft wrist restraints for at least 4 hours each will be included in the primary analysis.

SECONDARY OUTCOMES:
Sedation/Agitation | Baseline, every 60 minutes on study days 1-2, every 4 hours on study days 3-6
  Agitation will be measured via RASS (Richmond Agitation Sedation Scale) score. RASS is a validated and reliable ordinal measure of sedation/agitation status in the ICU ranging from -5 (extremely sedated, no response to voice or physical stimulation) to +4 (extremely agitated, violent, combative).
Delirium | Baseline, every 4 hours days 1-2, twice daily days 3-6
  Delirium will be measured via CAM-ICU (Confusion Assessment Method for the ICU). The CAM-ICU score is a validated and reliable binary measure of delirium status in the ICU. A "yes" score means delirium is present, and a "no score means delirium is absent.
Average cumulative dose of sedative medications | Up to 6 days
  Cumulative use of sedative medications over the 6 day study period
Average cumulative dose of analgesic medications | Up to 6 days
  Cumulative use of analgesics over the 6 day study period
Average cumulative dose of antipsychotic medications | Up to 6 days
  Cumulative use of antipsychotics over the 6 day study period

OTHER OUTCOMES:
Satisfaction with novel restraint (nurses, family, physicians, and patients when able) | Up to 6 days
  Satisfaction and acceptability will be assessed by the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) survey. The QUEST 2.0 is a valid, reliable, and widely used 12-question survey assessing satisfaction with technological devices. It is scored from 1-5, with >3.26 considered high satisfaction. The QUEST 2.0 has 2 subscales (satisfaction with device and with services). Satisfaction with the Exersides restraint will be assessed using the device subscale, which has good test-retest stability (ICC 0.82).
Acceptability of novel restraint (nurses, family, physicians, and patients when able) | Up to 6 days
  Acceptability will be assessed with semi-structured interviews using open-ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Renee Stapleton, MD, PhD, Principal Investigator — University of Vermont; Dale Needham, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - University of California San Diego, San Diego, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No